CLINICAL TRIAL: NCT02683382
Title: Effects of a Moisturizing Product on Dry Eye and Skin
Acronym: SDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petra Larmo (Industry)
Collaborators: Turun Silmäexpertit Oy, Turku, Finland (Unknown); Tekes - The Finnish Funding Agency for Technology and Innovation (Unknown); Finnsusp Oy, Lieto, Finland (Unknown)
Responsible Party: Sponsor-Investigator, Petra Larmo, Ph.D., R&D Manager, Aromtech Ltd.
Organization: Aromtech Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDE
Record Dates: First submitted 2016-02-02; First posted 2016-02-17 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moisturizing Eye Product (product in development) (Experimental): Moisturizing eye product in liquid form (medical device product in development). Part 1 of the study: Administered to both eyes 4 times/day for 1 day. Part 2: to one eye 4 times/day for 9 days. Part 3: to one eye 4 times/day for 45 days. Parts 2 & 3: treatment eyes randomized.
  Interventions: Device: Moisturizing Eye Product in Liquid Formula
- Moisturizing Eye Product, Comparison (Active Comparator): Moisturizing eye product in liquid form (medical device CE-marked). Part 2 of the study: Administered to one eye 4 times/day for 9 days. Treatment eyes randomized.
  Interventions: Device: Moisturizing Eye Product in Liquid Formula
- No treatment (No Intervention): Part 3 of the study: other eye is a control eye with no treatment for 45 days.

INTERVENTIONS:
Device: Moisturizing Eye Product in Liquid Formula — Moisturizing Eye Product in Liquid Formula for dry eyes and skin around the eyes
  Arms: Moisturizing Eye Product (product in development); Moisturizing Eye Product, Comparison

SUMMARY:
Dry eye is a common syndrome associated with symptoms of dryness, burning, itching and grittiness of eyes. The objective of this study is to investigate the effects of a moisturizing product in liquid formula on symptoms and signs of dry eye and on skin around the eyes.

ELIGIBILITY:
Inclusion Criteria:

* Dry eye symptoms OSDI score 20 or higher
* Dryness, burning or foreign body sensation moderate or higher

Exclusion Criteria:

* Severe eye diseases
* Known allergy to any of the ingredients of the product
* Laser surgery of eyes during the last year

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of dry eye: Ocular Surface Disease Index (OSDI), scores of dryness, burning and foreign body sensation of eyes | Part 1: baseline, 2, 4, and 6 hours. Part 2: baseline, 1 day, 3 and 9 days. Part 3: baseline and 45 days
Change in tear film osmolarity (mOsm/L) | Part 1: baseline, 2, 4, and 6 hours. Part 2: baseline, 1 day, 3 and 9 days. Part 3: baseline and 45 days
Change in tear film break-up time (s) | Part 1: baseline, 2, 4, and 6 hours. Part 2: baseline, 1 day, 3 and 9 days. Part 3: baseline and 45 days
Change in tear secretion, Schirmer test (mm/min) | Part 1: baseline, 2, 4, and 6 hours. Part 2: baseline, 1 day, 3 and 9 days. Part 3: baseline and 45 days
Change in signs of irritation of eyes, scoring by an eye specialist | Part 1: baseline, 2, 4, and 6 hours. Part 2: baseline, 1 day, 3 and 9 days. Part 3: baseline and 45 days
Change in transepidermal water loss from skin around the eyes (g/m2h) | Part 1: baseline, 2, 4, and 6 hours. Part 2: baseline, 1 day, 3 and 9 days. Part 3: baseline and 45 days

SECONDARY OUTCOMES:
Change in other symptoms of dry eye: soreness, grittiness, watery eyes, redness, blurring of eyes (daily symptom logbooks: scoring in scale from 0 to 3) | Part 2: change from baseline to 9 days; Part 3: change from baseline to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Minna Sandberg-Lall, MD, Principal Investigator — Turun Silmäexpertit Oy, Turku, Finland
Locations (1):
- Turun Silmäexpertit Oy, Turku, Finland

IPD SHARING:
Plan to Share IPD: No